CLINICAL TRIAL: NCT00505310
Title: Biobehavioral Effects of Emotional Expression in Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ID00-168; NCI-2012-02100 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Kidney Cancer
Keywords: Kidney Cancer; Renal Cell Carcinoma; Emotional Expression; Writing; Questionnaire; Survey
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Functional Laterality; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional Expression Writing (Experimental): 20 minutes of writing on different topics at four different times. Questionnaires about mood and quality of life completed 1 month, 4 months, and 10 months after the last writing assignment.
  Interventions: Behavioral: Writing; Behavioral: Questionnaire
- Neutral Writing (Experimental): 20 minutes of writing on different topics at four different times. Questionnaires about mood and quality of life completed 1 month, 4 months, and 10 months after the last writing assignment.
  Interventions: Behavioral: Writing; Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Writing — 20 minutes of writing on different topics at four different times.
Behavioral: Questionnaire — Questionnaires about mood and quality of life completed 1 month, 4 months, and 10 months after the last writing assignment.
  Other Names: Survey

SUMMARY:
The proposed study will assess the psychological and physiological benefits of an emotional expression intervention in patients with renal cancer. Patients will be randomly assigned to an emotional expression writing group or to a neutral writing group. This study will also evaluate the extent to which psychosocial factors mediate the intervention program and predict patients' recovery and adjustment to treatment. Potential mediators include level of cognitive processing, social networks/interactions, and sense of coherence and ability to find meaning in the illness experience.

Specific objectives of the proposed research are:

* To evaluate an emotional expression intervention in patients with renal cancer. Researchers will determine the extent to which an emotional expression writing-based intervention enhances adjustment during the first 12 months following diagnosis and treatment. Dimensions of adjustment will be assessed by examining indices of QOL, mental health, and stress (subjective symptoms of distress, perceived stress, and mood).
* To determine the effects of an emotional expression writing-based intervention on immune function. The immune measures assessed in this study will include both general and autologous tumor-specific immune responses including cytotoxicity to K562 target cells; cytotoxicity to autologous tumor target cells; and functional assessment of type-1 and type-2 cytokines using autologous tumor and polyclonal stimulants.
* To identify the psychosocial processes underlying the efficacy of the intervention.

DETAILED DESCRIPTION:
Patients in this study will already be scheduled for surgery/ablation, or for chemotherapy and/or radiation treatment. Patients undergoing surgery/ablation will complete some questionnaires about their mood and quality of life. These questionnaires will happen about 6 weeks after their procedure, during their scheduled visit to M.D. Anderson to follow-up after their surgery. Patients scheduled to receive chemotherapy and/or radiation treatment will complete the same questionnaires around the time of their new patient consult visit at M.D. Anderson. They should take about 60 minutes to complete. About 8 teaspoons of blood will be drawn to measure immune function.

Patients will then be randomly picked (as in the toss of a coin) to be in one of two groups. One group will be the emotional expression writing group. The other group will be the neutral writing group.

Patients in both groups will be asked to write for 20 minutes on different topics at four different times. They will be asked to complete all assignments in their home. They will choose four separate times when they would like to do the writing assignments and a research assistant will prompt them with a phone call at those times. During these phone calls, patients will complete a brief mood evaluation before the start of the writing session. After 20 minutes, patients will receive another phone call to signal that they should stop writing. A second mood assessment will also be given at this time. Patients will be provided with a pre-addressed, stamped envelope for mailing each writing sample back to M. D. Anderson the day after it is completed.

Patients will complete some questionnaires about their mood and quality of life approximately 1 month, 4 months, and 10 months after their last writing assignment. They should take about 60 minutes to complete. About 8 teaspoons of blood will then be taken each time to measure immune function.

This is an investigational study. As many as 710 patients will be enrolled in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1) Men or woman older than 18 years with stage I-IV renal cell carcinoma 2) Zubrod performance status of less than or equal to 2 3) have no serious intercurrent medical illness 4) read and speak English

Exclusion Criteria:

1) Score of 23 or below on the Mini-mental 2) History of primary or secondary immunodeficiency 3) Taking immunosuppressive drugs such as systemic corticosteroid 4) Patients who are undergoing a surgical procedure and do not sign the general tissue consent form 5) Patients with major psychiatric diagnoses or currently seeking psychological counseling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2002-08-21 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
To measure the psychological and physiological benefits of an emotional expression program in patients with kidney cancer. | 8 Years

SECONDARY OUTCOMES:
To learn how the expression of emotions affects quality of life, stress, and immune function. | 8 Years

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Snyder S, Milbury K, Wagner R, Cohen L. Words matter: The use of generic "you" in expressive writing in an oncology setting. J Health Psychol. 2024 Jan;29(1):42-51. doi: 10.1177/13591053231182218. Epub 2023 Jun 26. PMID 37358056
- [Derived] Milbury K, Spelman A, Wood C, Matin SF, Tannir N, Jonasch E, Pisters L, Wei Q, Cohen L. Randomized controlled trial of expressive writing for patients with renal cell carcinoma. J Clin Oncol. 2014 Mar 1;32(7):663-70. doi: 10.1200/JCO.2013.50.3532. Epub 2014 Jan 27. PMID 24470003
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org